CLINICAL TRIAL: NCT05337488
Title: Exploring the Contributing Factors of Solitary Drinking Among Hong Kong Chinese Adolescents and Young Adults
Brief Title: Contributing Factors of Solitary Drinking Among Adolescents and Young Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Other Study IDs: Solitary_drinking_1
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-04

CONDITIONS: Alcohol Drinking; Alcohol Use Disorder
MeSH Terms: conditions — Alcohol Drinking; Alcoholism | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject with solitary drinking behaviour: A convenience sample of 40 solitary drinkers aged between 10 and 24 will be invited to undergo complete a questionnaire and an individual semi-structured interviews.
  Interventions: Other: questionnaire with interview

INTERVENTIONS:
Other: questionnaire with interview — They will be invited to complete a questionnaire and an individual semi-structured interviews.

SUMMARY:
A convenience sample of 40 solitary drinkers aged between 10 and 24 will be invited to complete a structured questionnaire and a individual semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* 10-24 years old,
* able to speak Cantonese
* self-report as exhibiting solitary drinking behaviour

Exclusion Criteria:

* None

Ages: 10 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents and young adults with solitary drinking behaviour
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
solitary drinking episode | past 30 days
  assessed by a structured questionnaire
percent of drinking time spent on solitary drinking | past 30 days
  assessed by a structured questionnaire

IPD SHARING:
Plan to Share IPD: No